CLINICAL TRIAL: NCT01635777
Title: Safety and Efficacy of Oral Miltefosine in Patients With Post Kala Azar Dermal Leishmaniasis (PKDL)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AB Foundation (Other)
Collaborators: World Health Organization (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Z015
Record Dates: First submitted 2012-07-03; First posted 2012-07-10 (Estimated); Last update posted 2012-07-10 (Estimated); Status verified 2012-07

CONDITIONS: PKDL
Keywords: PKDL; miltefosine
MeSH Terms: interventions — miltefosine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 12 weeks (Experimental): miltefosine 12 weeks
  Interventions: Drug: Miltefosine
- 8 weeks (Experimental): miltefosine 8 weeks
  Interventions: Drug: Miltefosine

INTERVENTIONS:
Drug: Miltefosine — 2.5 mg/kg/day for 12 weeks
  Arms: 12 weeks
Drug: Miltefosine — 2.5 mg/kg/day for 8 weeks
  Arms: 8 weeks

SUMMARY:
Miltefosine efficacy will be >85%

ELIGIBILITY:
Inclusion Criteria:

* 12 years or older
* nodules and papules consistent with post kala-azar dermal leishmaniasis
* parasitological confirmation of Leishmania infection

Exclusion Criteria:

* platelet count <100x 109/l,
* leukocyte count <2.5 x 109/l ,
* hemoglobin < 8.0 g/100 ml ,
* liver function tests >3 times upper limit of normal range,
* bilirubin >2 times upper limit of normal range,
* serum creatinine or blood urea nitrogen >1.5 times upper limit of normal range);
* any non-compensated or uncontrolled condition,
* lactation, pregnancy, or likelihood of inadequate contraception in females of childbearing potential for the treatment period plus 2 months thereafter;
* treatment with any anti-leishmanial drug within the previous 12 weeks.

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2007-07; Primary Completion 2009-10 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Cure rate | 12 months after end of treatment

SECONDARY OUTCOMES:
adverse events | during therapy: the 8 weeks of therapy for the 8 week treatment group and 12 weeks of therapy for the 12 week treatment group
  gastrointestinal events: vomiting and diarrhea

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Medical Sciences, Banaras Hindu University,, Varanasi, India